CLINICAL TRIAL: NCT00957164
Title: Treatment of PTSD and Chronic Pain After Traumatic Orthopedic Injury: A Randomized Clinical Trial
Brief Title: Treatment of Post-Traumatic Stress Disorder (PTSD) and Chronic Pain After Traumatic Orthopedic Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Collaborators: 59th Medical Wing (U.S. Federal Agency); Brooke Army Medical Center (U.S. Federal Agency); The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STRONGSTAR*PAIN*PTSD
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Pain; Post-traumatic Stress Disorder
Keywords: Chronic pain; PTSD
MeSH Terms: conditions — Chronic Pain; Stress Disorders, Post-Traumatic | interventions — Self Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pain Treatment Only (Active Comparator): Pain treatment will involve five-sessions over 5 weeks of individual treatment protocol based on the existing chronic pain management program through the Clinical Health Psychology Service at Wilford Hall Medical Center. This treatment will involve covering the difference between chronic and acute pain, the role of cognitive, behavioral, and emotional variables in pain progression, and ways to manage these variables to prevent the development of chronic pain.
  Interventions: Behavioral: Chronic Pain Management Treatment; Behavioral: Self-Care
- PTSD Treatment Only (Active Comparator): The PTSD treatment used in this study is an adaptation of a brief Prolonged Exposure treatment protocol for PTSD as illustrated in a 2005 paper published by Cigrang, Peterson, and Schobitz in which a 4-session prolonged exposure treatment was used to address PTSD symptoms in three injured soldiers recently exposed to trauma. The authors found a 50+% decrease in PTSD symptoms after these four sessions. The present study will rely upon a similar brief PTSD intervention for treating chronic PTSD among trauma-exposed injured active duty service members. The PTSD intervention will be expanded into five sessions over 5 weeks to include an initial session for assessment and education on the co-morbidity of pain and PTSD. All PTSD treatment will be provided under the direct care or supervision of a Master Trained therapist in Prolonged Exposure.
  Interventions: Behavioral: Brief Prolonged Exposure Protocol; Behavioral: Self-Care
- Combined Pain and PTSD Treatment (Active Comparator): This treatment arm will involve 5 sessions each of the Pain-Only and PTSD-Only treatments described above.
  Interventions: Behavioral: Brief Prolonged Exposure Protocol; Behavioral: Chronic Pain Management Treatment
- Treatment as Usual (No Intervention): The treatment as usual group will complete the assessments given in each of the other study arms, but will not participate in treatment through the study. Instead, participants randomized to this group will be encouraged to seek treatment for pain and/or PTSD through existing channels. Referrals for treatment will be made for those with clinically significant symptoms for pain and/or PTSD at intake.

INTERVENTIONS:
Behavioral: Brief Prolonged Exposure Protocol — The PTSD treatment used in this study is an adaptation of a brief Prolonged Exposure treatment protocol for PTSD as illustrated in a 2005 paper published by Cigrang, Peterson, and Schobitz 54 in which a 4-session prolonged exposure treatment was used to address PTSD symptoms in three injured soldiers recently exposed to trauma. The authors found a 50+% decrease in PTSD symptoms after these four sessions. The present study will rely upon a similar brief PTSD intervention for treating chronic PTSD among trauma-exposed injured active duty service members. The PTSD intervention will be expanded into five sessions over 5 weeks to include an initial session for assessment and education on the co-morbidity of pain and PTSD. All PTSD treatment will be provided under the direct care or supervision of a Master Trained therapist in Prolonged Exposure.
  Arms: Combined Pain and PTSD Treatment; PTSD Treatment Only
Behavioral: Chronic Pain Management Treatment — Pain treatment will involve five-sessions over 5 weeks of individual treatment protocol based on the existing chronic pain management program through the Clinical Health Psychology Service at Wilford Hall Medical Center. This treatment will involve covering the difference between chronic and acute pain, the role of cognitive, behavioral, and emotional variables in pain progression, and ways to manage these variables to prevent the development of chronic pain.
  Arms: Combined Pain and PTSD Treatment; Pain Treatment Only
Behavioral: Self-Care — participants randomized to either the Pain-only or PTSD-only groups will receive five sessions of pain- or PTSD-specific treatment followed by five sessions of self-care placebo over 5 weeks. The self-care module will be manualized for reliability and fidelity between providers and will involve 60-minute sessions covering various topics.
  Arms: PTSD Treatment Only; Pain Treatment Only

SUMMARY:
The purpose of this study is to examine the efficacy of multiple treatment options in addressing the co-morbidity between pain and PTSD symptoms. Recent research has suggested that pain and PTSD co-morbidity presents unique problems for pain and PTSD treatment, and new approaches are desperately needed to address this issue. To this end, the investigators hope to identify the efficacy of a combined pain and PTSD psychosocial treatment protocol compared to that of stand-alone psychosocial treatments for pain and PTSD. The primary measure for treatment efficacy will be treatment-related changes in measures of psychosocial and functional outcomes associated with chronic pain and PTSD conditions. The investigators will additionally measure socioeconomic outcomes including return to pre-trauma job (or a job of similar capacity), maintenance of active duty work at pre-trauma capacity for 6 and/or 12 months after return, and number of healthcare appointments made between follow-ups for pain or PTSD treatment.

DETAILED DESCRIPTION:
This study will use a four-group randomized experimental design similar to that used in a study currently being conducted by John Otis with VA patients with chronic pain/chronic PTSD. The four groups will include Pain Treatment (PAIN) only, PTSD Treatment (PTSD) only, Pain and PTSD Treatments (PAIN+PTSD), and treatment as usual (TAU). The investigators hypothesize that treating individuals with chronic pain and PTSD (e.g., more than 6 months in duration) symptoms through a proven psychosocial model will help to improve psychological, socioeconomic and physical symptoms of these chronic clinical syndromes that have been shown to be unfortunately recalcitrant to treatment and enormously costly both to society healthcare and, more importantly, to the person suffering from enduring pain and traumatic stress. We further hope to demonstrate the efficacy of these early treatments in facilitating the return to active duty of military personnel suffering from pain and traumatic stress. Finally, we hope to positively impact other psychosocial and socioeconomic outcomes such as work retention (as measured by self-report work status and retention of work at 6- and 12-month follow-up), additional health-care utilization (as measured by self-report of number of PTSD or pain-related healthcare visits), depression symptoms (as measured by the Beck Depression Inventory), health-related quality of life (as measured by the SF-36), and perceived disability (as measured by the Million Visual Analog Scale). Evaluations of these four groups will be conducted at pre-treatment, immediately at the post-treatment, and at 6- and 12-month follow-up periods in order to determine differential outcomes on variables such as PTSD and pain symptom presence/severity, self-reported pain and disability, functional gains, satisfaction with treatment, return to active duty, retention of pre-trauma work capacity at 6- and 12-month follow-up, and additional health-care utilization as measured by number of healthcare appointments attended for pain or PTSD symptom management. The initial post-treatment evaluation will occur at the end of the ten-week treatment interval for each individual's randomization block. For those in the treatment as usual (TAU) group, post-treatment assessment will occur ten weeks after pre-treatment assessment is completed. Changes in functional activity status, psychosocial functioning, and satisfaction with treatment will also be systematically evaluated before, immediately after, and during the post-treatment periods. It should be noted that many of the PAIN-only, and TAU subjects may receive some type of standard care for PTSD symptoms if they access those services on their own. The same could be true for the PTSD-only and TAU subjects. They may also receive some type of standard care for pain symptoms that they access on their own. The investigators will monitor any such services received in order to attempt to control for possible spurious effects of outside treatment in later analyses.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* hospital admission for any traumatic orthopedic injury defined as any musculo-skeletal injury requiring convalescence and/or surgery that is deployment related.
* Fluency in English
* Glasgow Coma Score (GCS) = 15 at time of hospital discharge
* willingness and ability to meet study follow-up requirements
* PTSD CheckList - Military (PCL-M) > 30
* duration of any amount of pain >12 weeks based on self-report and date of injury, and PTSD symptoms of > to 4 weeks.
* Pain Disability Questionnaire (PDQ) > 30
* no current need for surgical intervention for pain
* be stable on any psychotropic medications they may be taking. (Participants will be required to meet psychotropic medication stabilization criteria for the periods preceding and overlapping with the diagnostic assessment and treatment. This criterion is established in order to minimize the likelihood that significant outcome effects may be attributed to changes in psychotropic medications rather than to the treatment protocol.)
* medically cleared for study participation by Orthopedic provider or collaborating study physician
* Active Duty Military, Reserve, or Activated Reservist

Exclusion Criteria:

* head injury greater than mild TBI as assessed by an inability to consent to the study and complete the baseline psychological testing
* current pregnancy will exclude participation in Functional Capacity Evaluation (FCE) assessment, but not study participation. Pregnancy will be assessed by self-report
* current diagnosis of schizophrenia, bipolar disorder, or other psychotic disorder as identified by clinical interview
* primary diagnosis of burn injury, though burn patients will be eligible if burn is a secondary diagnosis and not the primary reason for pain
* participant is currently taking a benzodiazepine medication for PTSD symptoms
* unstable suicidal ideation
* currently receiving prolonged exposure treatment for PTSD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-08; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Post Traumatic Stress Disorder Symptoms/Diagnosis | 1 Year
Chronic Pain Intensity | 1 Year
Self-reported disability | 1 Year

SECONDARY OUTCOMES:
Depression/Suicidality | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Gatchel, Ph.D., Principal Investigator — University of Texas at Arlington; Donald D. McGeary, Ph.D., Principal Investigator — Wilford Hall Medical Center, USAF; Mysti R. Moore, MPT, Study Director — University of Texas at Arlington
Locations (4):
- United States (4):
  - The University of Texas at Arlington, Arlington, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas